CLINICAL TRIAL: NCT01787279
Title: Expanded Access Programme of PEGASYS® (Peg Interferon Alpha-2a 40KD) in Patients With HBe-Ag-negative Chronic Hepatitis B
Brief Title: An Expanded Access Study of Pegasys (Peginterferon Alfa-2a) in Patients With HBeAg-Negative Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19522
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (1):
- Peginterferon alpha-2a, 180 mcg/48 weeks (Experimental): Eligible participants with HI3vAg (a type of Hepatitis B surface antigen) negative chronic hepatitis B will be administered peginterferon alpha-2a (PEGASYS), 40kD, 180 micrograms (mcg) subcutaneously once weekly for 48 weeks. The untreated Follow-up will be for 24 weeks.
  Interventions: Drug: Peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: Peginterferon alfa-2a [Pegasys] — 180 mcg subcutaneously weekly, 48 weeks

SUMMARY:
This is an expanded access programme to make Pegasys (peginterferon alfa-2a) available to patients with HBeAg-negative chronic hepatitis B in Morocco. Patients will receive Pegasys 180 mcg subcutaneously weekly for 48 weeks and efficacy and safety will be recorded during treatment and for 24 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 and </= 70 years of age
* HBeAg-negative chronic hepatitis B
* HBsAg-positive for at least 6 months, anti- hepatitis B (HBs) negative
* Serum alanine transaminase (ALT) > 2 ULN (upper limit of normal) but </= 10 x Upper limit of normal (ULN)
* Hepatitis B virus (HBV) DNA > 10'000 copies/ml (Roche Monitor or Taqman)
* No previous treatment with interferon (standard or pegylated) or with a nucleoside analogue
* Women of childbearing potential must agree to use reliable contraception during the study and for 3 months after treatment completion

Exclusion Criteria:

* Previous antiviral interferon-based therapy for chronic hepatitis B
* Pregnant and lactating women
* Evidence of decompensated liver disease
* Co-infection with active hepatitis A, hepatitis C, hepatitis D and/or human immunodeficiency virus (HIV)
* History or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis
* Previous or current hepatocellular carcinoma
* History or other evidence of bleeding from oesophageal varices or other conditions consistent with decompensated liver disease
* Inadequate hematologic or renal function
* Serum bilirubin level > 2 times the upper limit of normal
* Severe psychiatric disease
* History of severe seizure disorder or current anticonvulsant use
* History of evidence of any disease or condition which would make the patient, in the opinion of the investigator, unsuitable for the study
* Evidence of drug abuse within one year of study entry
* Alcohol intake of more than 3 standard drinks per day for men and 2 standard drinks per day for women (1 standard drink contains 10 g of alcohol)
* Participation in another trial or receipt of an investigational drug within 12 weeks prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Morocco (2):
  - Casablanca
  - Rabat

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 59 participants were enrolled in this study conducted from 13 January 2006 to 25 May 2009 at 9 centers in Kingdom of Morocco.
Groups:
- Peginterferon Alpha-2a, 180 mcg/48 Weeks: Eligible participants with HI3vAg (a type of hepatitis B surface antigen) negative chronic hepatitis B administered peg interferon alpha-2a (PEGASYS), 40 kilodalton (kD), 180 micrograms (mcg), subcutaneously, once weekly for 48 weeks. The untreated follow-up was for 24 weeks.
Period: Overall Study
Arm/Group | Peginterferon Alpha-2a, 180 mcg/48 Weeks
Started | 59
Completed | 56
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all the participants who received at least one dose of study medication and have one subsequent post baseline safety assessment
Groups:
- Peginterferon Alpha-2a, 180 mcg/48 Weeks: Eligible participants with HI3vAg (a type of hepatitis B surface antigen) negative chronic hepatitis B administered PEGASYS, 40kD, 180 mcg, subcutaneously once weekly for 48 weeks. The untreated follow-up was for 24 weeks.
Arm/Group | Peginterferon Alpha-2a, 180 mcg/48 Weeks
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hepatitis C Virus Deoxyribonucleic Acid <10,000 Copies/Milliliter at Week 72
Description: Participants who had Hepatitis B Virus Deoxyribonucleic Acid (HBV-DNA) levels below 100,000 copies per milliliter (mL) at the end of follow-up (at Week 72) were reported.
Time Frame: At Week 72
Population: Intent-to-treat (ITT) population included all the participants who received at least one dose of study medication and had one subsequent post baseline assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alpha-2a, 180 mcg/48 Weeks
Number analyzed (Participants) | 59
Percentage of participants | 65.4 [52.5 to 78.3]

2. Primary Outcome: Percentage of Participants Achieving Normalization of Alanine Aminotransferase at Week 72
Description: Percentage of participants with a normal serum alanine aminotransferase (ALT) level at the end of the study was analyzed. Normal ranges for ALT are 7 to 56 International Units/Litre. Participants with ALT less than the upper limit of normal at end of treatment were reported.
Time Frame: At Week 72
Population: ITT population included all the participants who received at least one dose of study medication and had one subsequent post baseline assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alpha-2a, 180 mcg/48 Weeks
Number analyzed (Participants) | 59
Percentage of participants | 68.6 [56.8 to 80.4]

3. Primary Outcome: Number of Participants With Any Adverse Events and Serious Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. A serious adverse event (SAE) is any significant hazard, contraindication, side effect that is fatal or life-threatening, requires hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability/ incapacity, is a congenital anomaly/ birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above
Time Frame: Up to Week 72
Population: Safety analysis population is defined to include only participants who receive at least one dose of study medication and have one subsequent post baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alpha-2a, 180 mcg/48 Weeks
Number analyzed (Participants) | 59
Participants
  Any AE | 46
  Any SAE | 0

4. Secondary Outcome: Percentage of Participants Achieving Hepatitis B Virus DNA < 400 Copies/mL at Week 72
Description: Participants who had HBV-DNA levels below 400 Copies/mL at the end of follow-up (at Week 72) were reported.
Time Frame: At Week 72
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alpha-2a, 180 mcg/48 Weeks
Number analyzed (Participants) | 59
Percentage of participants | 26.9 [14.8 to 39.0]

5. Secondary Outcome: Percentage of Participants Achieving Hepatitis B Surface Antigen Seroconversion at Screening and Week 48
Description: Seroconversion is defined as the absence of hepatitis B surface antigen (HBsAg) with a negative result for HBsAg and the presence of anti-Haemoglobin (HBs) antibodies (a positive result for anti-HBs) determined at Week 48. Blood samples were analyzed to check whether it is HBsAg-negative and anti-HBs antibodies positive.
Time Frame: At Screening and Week 48
Population: ITT population included all the participants who received at least one dose of study medication and had one subsequent post baseline assessment. 'n'=number of evaluable participants available at specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Peginterferon Alpha-2a, 180 mcg/48 Weeks
Number analyzed (Participants) | 59
Percentage of participants
  HBs-Ag Negative, Screening (n= 59) | 1.7
  HBs-Ag Negative, Week 48 (n= 55) | 10.9
  Anti-HBs Positive, Screening (n= 59) | 0
  Anti-HBs Positive, Week 48 (n= 55) | 10.9

6. Secondary Outcome: Percentage of Participants Achieving Combined Response Hepatitis B Virus DNA < 10,000 Copies/mL and Normal ALT at Week 72
Description: Percentage of participants showing normal ALT values and HBV DNA levels <10,000 copies/ mL were reported.
Time Frame: At Week 72
Population: ITT population included all the participants who received at least one dose of study medication and had one subsequent post baseline assessment. Participants available at the time of assessment were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Peginterferon Alpha-2a, 180 mcg/48 Weeks
Number analyzed (Participants) | 51
Percentage of participants | 58.8

ADVERSE EVENTS:
Time Frame: Up to Week 72
Description: An AE is any untoward medical occurrence in a participant or clinical investigation that does not necessarily have to have a causal relationship with treatment. An AE can be unfavourable and unintended sign, symptom, or disease associated with a medicinal product, whether or not considered related to the medicinal product.
Groups:
- Peginterferon Alpha-2a, 180 mcg/ 48 Weeks: Eligible participants with HI3vAg (a type of hepatitis B surface antigen) negative chronic hepatitis B administered PEGASYS, 40kD, 180 mcg, subcutaneously once weekly for 48 weeks. The untreated follow-up was for 24 weeks.
Arm/Group | Peginterferon Alpha-2a, 180 mcg/ 48 Weeks
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 40/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alpha-2a, 180 mcg/ 48 Weeks (N=59)
Asthenia (General disorders) | 23
Arthralgia (General disorders) | 4
Anxiety (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights